CLINICAL TRIAL: NCT04120558
Title: Comparing OutcomeS of Through Knee and Above Knee Amputation (COSTAA)
Brief Title: Comparing OutcomeS of Through Knee and Above Knee Amputation
Acronym: COSTAA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: R2378
Record Dates: First submitted 2019-09-26; First posted 2019-10-09 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Through Knee Amputation
MeSH Terms: interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Through knee amputees: Community dwelling individuals with through knee amputation of all mobility levels.
  Interventions: Other: Qualitative interviews and focus groups; Other: Functional mobility tests and questionnaires
- Above knee amputees: Community dwelling individuals with above knee amputation of all mobility levels.
  Interventions: Other: Qualitative interviews and focus groups; Other: Functional mobility tests and questionnaires

INTERVENTIONS:
Other: Qualitative interviews and focus groups — Semi-structured interviews will be undertaken with at least 24 and up to as many as 36 through knee and above knee amputees. A topic guide will be used to interview participants about perceived functional ability, body image, adapting post amputation and overall quality of life. A sampling frame will be used to ensure a range of views are sought (e.g. both men and women with through and above knee amputations; and with different mobility levels). Thematic analysis will be used to analyse the data. Focus group discussions will be informed by the findings of the interviews.
  The themes that emerge from the semi-structured interviews will be further explored using focus groups and allow for comparison of the experiences between through knee and above knee amputees.
Other: Functional mobility tests and questionnaires — Function in sitting and sit-and-reach will be assessed in non-ambulatory (wheelchair users) individuals. An overall score for each sitting activity will be recorded and the distance reached will be calculated.
  Walking, timed-up-and-go, L-test, balance in sitting and standing, seated activities will be assessed in ambulatory (prosthetic using) individuals. The time taken, distance walked, distance reached, and the overall scores for each activity will be compared between the two groups. Fear of falls and confidence levels when performing tasks will be investigated using two questionnaires.
  The EQ-5D-5L and SF-36 will be issued to the non-ambulatory and ambulatory participants to complete when attending the testing session.
  The Locomotor Capability Index - 5 (LCI-5), Activities-specific Balance Confidence Scale (ABC-UK) and Houghton scale of prosthetic use in people with lower-extremity amputations

SUMMARY:
Major lower limb amputation is a life changing surgical procedure to treat complications of diabetes mellitus and peripheral vascular disease. The level of function after amputation is dependent on pre-morbid levels of activity, age, co-morbidities and the level of amputation. The level of amputation performed is determined by level of disease and surgical assessment. Below knee amputation provides the best functional outcomes due to the benefits of keeping the knee intact. When a below knee amputation is not possible, routine practice is to perform an above knee amputation. Greater challenges for rehabilitation present at this level due to the shorter lever. Amputation through the knee is less commonly performed despite its reported benefits which include a long mechanical lever arm, an endbearing stump and greater muscle control.

A recent systematic review recommends further comparison of through knee and above knee amputation. The recommended areas of research are gait biomechanics and quality of life for these patient groups. Therefore, the aim of this research is to compare and contrast the long-term functional mobility and quality of life outcomes of limb wearing through knee and above knee amputees. The study will be split into two workstreams, the first focusing on functional outcomes and the second focusing on quality of life using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling adults aged 18 or over.
* People who have had either a through-knee or above-knee amputation.
* Unilateral amputees.
* English speaking and cognitively be able to follow instructions and fill out questionnaires independently.

Exclusion Criteria:

* People are unable to provide an informed consent.
* People who have a below-knee amputation.
* Unable to transfer with assistance of one.
* Unable to walk more than 5 metres (ambulatory section workstream 1 only).
* Individuals will be excluded from workstream 2 if they report another health condition with greater impact on their quality of life than their amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults with through knee or above knee amputation of all mobility levels.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes measure for workstream 1 is walking speed. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Walking speed will be determined as distance divided by time in seconds and will be calculated during timed-up-and-go test, L-test, two-minute walk test (2MWT) and six-minute walk test (6MWT). The results will be presented as metres per second
The primary outcome measure for workstream 2 is an in-depth analysis and comparison of quality of life. | Through study completion, an average of 1 year
  The analysis of semi-structured interviews and focus groups using a self designed topic guide with questions relating to quality of life.

SECONDARY OUTCOMES:
The secondary outcome measures for workstream 1 include time taken. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Time taken will be calculated as the time in seconds calculated during timed-up-and-go test and L-test.
The secondary outcome measures for workstream 1 include distance reached. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Distance reached will be calculated as the distance reached in centimetres calculated during the functional reach test, and the sit-and-reach test.
The secondary outcome measures for workstream 1 include distance walked. [ | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Distance walked will be calculated as the distance in metres calculated during the 2MWT and 6MWT.
The secondary outcome measures for workstream 1 include step count. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Step count will be calculated as the number of steps taken during timed-up-and-go test, L-test, 2MWT and 6MWT.
The secondary outcome measures for workstream 1 include predicted 6MWT score. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Predicted 6MWT score will be calculated as the distance walked in the 2MWT multiplied by 3.
The secondary outcome measures for workstream 1 include time taken to stand from sitting. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  The time taken to stand from sitting will be calculated as the time in seconds taken from the participant moving from a seated to standing position. This will be calculated during the Timed-Up-and-Go test and the L-test.
The secondary outcome measures for workstream 1 include time taken to sit from standing. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  The time taken to sit from standing will be calculated as the time in seconds taken from the participant moving from a standing to seated position. This will be calculated during the Timed-Up-and-Go test and the L-test.
The secondary outcome measures for workstream 1 include walking time. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  The walking time will be calculated as the time in seconds spent walking to and from the chair. This will be calculated during the Timed-Up-and-Go test and the L-test.
The secondary outcome measures for workstream 1 include functional balance. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Functional balance will be calculated as the overall score from their observed performance across 14 activities when completing the Berg Balance scale.
The secondary outcome measures for workstream 1 include function during sitting. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Function during sitting will be calculated as the overall score from their observed performance across 14 activities when completing the function in sitting test.
The secondary outcome measures for workstream 1 include step length and height. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Step length and height will be observed and recorded as part of the Tinetti assessment.
The secondary outcome measures for workstream 1 include step symmetry. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Step symmetry will be observed and recorded as part of the Tinetti assessment.
The secondary outcome measures for workstream 1 include falls risk using the Tinetti assessment. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Falls risk will be calculated as the overall score from their observed performance out of 28 when completing the Tinetti assessment.
The secondary outcome measures for workstream 1 include recording of confidence levels using the Activity Balance Confidence (ABC-UK) questionnaire. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Confidence levels will be calculated using the Activity-Balance Confidence (ABC-UK) questionnaire.
  Items are rated on a scale 0-100, 0 represents no confidence and 100 represents complete confidence when performing activities.
The secondary outcome measures for workstream 1 include confidence levels using the Locomotor-Capabilities Index-5 (LCI-5) questionnaire. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Confidence levels will be calculated using the Locomotor-Capabilities Index-5 (LCI-5) questionnaire. Items are scored on a 4 point scale ranging from 0 = not able to accomplish activity alone 3= being able to accomplish the activity alone.
The secondary outcome measures for workstream 1 include confidence levels using the Short Form Survey Instrument (SF36) | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Confidence levels will be calculated using the Short Form Survey Instrument (SF36). Items are scored using Likert scale and yes/no options. Scales are standardised with a scoring algorithm to obtain a score ranging from 0-100. High scores indicate better health status.
The secondary outcome measures for workstream 1 include confidence levels using Houghton's Scale of Prosthetic Use. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Confidence levels will be calculated using Houghton's Scale of Prosthetic Use. This is a 4 item instrument to capture prosthetic wearing habits. Users will have a total score out of 12 where a high score indicates great performance and great comfort. The first 3 items are scored on a 4 point scale ranging from 0-3 where 0=low level of confidence and 3 = high level of confidence. The 4th item is a yes/no question relating to stability where yes scores 0 and No scores 1.
The secondary outcome measures for workstream 1 include confidence levels using the EuroQol EQ-5D-5L questionnaire. | Measures taken at baseline visit, data reported through study completion, an average of 1 year
  Confidence levels will be calculated using the EQ-5D-5L questionnaire. EQ-5D-5L is a standardized instrument for measuring generic health and mobility. Scores are calculated using a likert scale 1-5 to indicate levels of severity where 1 = no problems and 5 = high level of problems. The EQ-5D-5L also includes a Visual Analogue Scale (EQ-VAS) score, users rate their perception of their health on a scale of 0-100 where 0=worst and 100=best health.
The secondary outcome measures for workstream 2 are the lived experiences, processes of adjustment, body image, satisfaction with prosthesis and overall quality of life differences between the through knee and above knee amputees. | Through study completion, an average of 1 year
  The analysis of semi-structured interviews and focus groups using a topic guide with self-designed questions relating to the lived experiences, processes of adjustment, body image, satisfaction with prosthesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, East Riding Of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No